CLINICAL TRIAL: NCT07369037
Title: Association of Prognostic Nutritional Index and Controlling Nutritional Status Score With 2-Year Clinical Outcomes in Patients With ST Elevation Myocardial Infarction
Brief Title: Association of Prognostic Nutritional Index and Controlling Nutritional Status Score With ST Elevation Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, OGUZHAN CELIK, Associate Professor, Muğla Sıtkı Koçman University
Other Study IDs: muglaSKU-CRD-OC-03
Record Dates: First submitted 2026-01-18; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: CONUT Score; ST Elevation (STEMI) Myocardial Infarction; Mortality
Keywords: conut score; pni score; ST Elevation (STEMI) Myocardial Infarction; mortality; quality of life
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
It is well known that malnutrition is a prognostic risk factor in chronic heart failure (CHF). Weight loss and the development of cardiac cachexia are associated with poor prognosis in CHF. However, objective indices such as the Prognostic Nutrition Index (PNI) and Controlling Nutritional Status (CONUT) have been developed and are widely used today to assess nutritional status. The CONUT index is an effective scoring system for monitoring pre- and post-hospital malnutrition status and is measured by serum albumin level, total cholesterol (TC), and lymphocyte count. PNI, calculated from serum albumin level and lymphocyte count, is another formula reflecting nutritional status and is well known to be associated with the risk of perioperative complications, especially in surgical patients. Only simple blood biomarkers are required to determine these two indices. The aim of this study is to evaluate the effect of nutritional status at admission, assessed by two objective nutritional indices, CONUT and PNI, on the outcomes of STEMI (ST elevation myocardial infarction) patients during a median follow-up period of two years.

DETAILED DESCRIPTION:
The prognostic impact of nutritional status in cardiovascular disease (CVD) is not fully understood. Clinical studies have shown that low serum albumin levels are associated with an increased risk of heart failure. Similarly, particularly in recent studies, hypoalbuminemia at hospital admission has been shown to independently predict long-term mortality in patients with ST-elevation myocardial infarction (STEMI) undergoing primary percutaneous coronary intervention. Malnutrition is well-known to be a prognostic risk factor in chronic heart failure (CHF). Weight loss and the development of cardiac cachexia are associated with poor prognosis in CHF. However, objective indices such as the Prognostic Nutrition Index (PNI) and Controlling Nutritional Status (CONUT) have been developed and are widely used today to assess nutritional status. The CONUT index is an effective scoring system for monitoring pre- and post-hospital malnutrition status and is measured by serum albumin level, total cholesterol (TC), and lymphocyte count. PNI, calculated using serum albumin level and lymphocyte count, is another formula reflecting nutritional status and is well-known to be associated with the risk of perioperative complications, especially in surgical patients. Only simple blood biomarkers are required to determine these two indices.

The aim of this study is to evaluate the effect of nutritional status at admission, assessed by two objective nutritional indices, CONUT and PNI, on the outcomes of STEMI patients during a median follow-up period of two years.

Variables will be expressed as frequency, mean, and standard deviation, and patients will be categorized according to their CONUT score (low ≤ 2 - high ≥ 3) and PNI score (PNI ≥ 45 and PNI < 45). The Pearson Chi-square test will be used to investigate whether there are differences between subgroups in terms of CONUT and PNI scores. If a normal distribution is observed for continuous variables, a Student t-test will be performed to determine the difference between groups. The method planned was to retrospectively analyze all consecutive patients diagnosed with STEMI who underwent primary percutaneous coronary intervention at three different centers (Muğla Training and Research Hospital Cardiology Clinic, Eskişehir City Hospital Cardiology Clinic, and Eskişehir Osmangazi Faculty of Medicine Cardiology Clinic). Laboratory, ECG, and echocardiographic findings at admission, as well as in-hospital and long-term outcomes, were planned to be monitored from patient files.

ELIGIBILITY:
Inclusion Criteria:

* All patients over 18 years of age diagnosed with ST-elevation myocardial infarction (STEMI) treated percutaneously within the specified date range.

Exclusion Criteria:

* Patients under 18 years of age Patients for whom laboratory data is unavailable Patients with incomplete data Patients diagnosed with cancer Patients with hematological diseases Patients using glucocorticoid drugs Patients with liver disease Patients with kidney disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A retrospective analysis of all major sequential calculations in 18 stages of past ST-elevation myocardial infarction (STEMI) diagnoses was planned. The analysis would examine disease-triggering factors, laboratory findings at admission, ECG and echocardiographic findings, as well as distribution, in-hospital, and long-term outcomes.
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Relationship between CONUT score and PNI index and mortality | 2 years
  The aim of this study is to evaluate the impact of nutritional status at admission, assessed by two objective nutritional indices, CONUT and PNI, on outcomes in STEMI patients during a median follow-up period of two years.Patients will be categorized according to their CONUT score (low ≤ 2 - high ≥ 3) and PNI score (PNI ≥ 45 and PNI < 45). The relationship between CONUT and PNI scores and mortality will be investigated.

CONTACTS AND LOCATIONS:
Locations (1):
- Mugla Sitki Kocman University, Menteşe, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No